CLINICAL TRIAL: NCT05952570
Title: The Impact of Predialytic Oral Protein-based Supplements on Nutritional Status and Quality of Life in Hemodialysis Patients
Brief Title: Impact of Predialytic Oral Protein on Nutritional Status and Quality of Life in HD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mohamed Mamdouh Mahmoud Mohamed Elsayed , MD, Lecturer, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: oral protein in HD
Record Dates: First submitted 2023-07-02; First posted 2023-07-19 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Hemodialysis Complication
Keywords: oral protein; Protein Supplementation; Hemodialysis; quality of life

STUDY DESIGN:
Intervention Model Description: This research is a randomized multi-center clinical trial in which 100 hemodialysis patients will be randomly assigned to one of the study groups using block randomization with a ratio of 1:1.
  * Group A: 50 patients will receive oral protein nutritional supplement (Fresubin protein powder 25mg/5scoops per hemodialysis session) 1 hour before the start of the session (predialytic) for 3 months.
  * Group B: 50 patients will receive a routine nutrition regimen for 3 months. (control group)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- protein supplement (Experimental): 50 patients will receive oral protein nutritional supplement (Fresubin protein powder 25mg/5scoops per hemodialysis session) 1 hour before the start of the session (predialytic) for 3 months
  Interventions: Dietary Supplement: oral protein nutritional supplement (Fresubin protein powder)
- control (Placebo Comparator): 50 patients will receive a routine nutrition regimen for 3 months. (control group)
  Interventions: Other: routine nutrition regimen

INTERVENTIONS:
Dietary Supplement: oral protein nutritional supplement (Fresubin protein powder) — 50 patients will receive oral protein nutritional supplement (Fresubin protein powder 25mg/5scoops per hemodialysis session) 1 hour before the start of the session (predialytic) for 3 months
  Arms: protein supplement
Other: routine nutrition regimen — 50 patients will receive a routine nutrition regimen for 3 months. (control group)
  Arms: control

SUMMARY:
The aim of this work is to study the effects of oral protein-based supplements on nutritional status in hemodialysis patients

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a prevalent chronic condition and the incidence of end-stage renal disease (ESRD) is expected to increase over the next few decades. In patients with CKD, especially in those with ESRD and undergoing maintenance dialysis therapy (MDT), a state of metabolic and nutritional derangements, more aptly called protein-energy wasting (PEW), caused by a combination of insufficient intake, uremic toxins, inflammation, and superimposed catabolism, plays a major role among the many risk factors that affect outcomes of CKD .

Oral nutritional supplement (ONS) is a simple and effective way to supplement energy and protein to malnourished patients on the basis of regular diet. Therefore, if the protein of regular diet in dialysis patients are not enough, they should be supplemented with (ONS) when appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Adult hemodialysis patients (≥18 years of age).
* Received dialysis for at least 6 months prior to study screening.
* Receive hemodialysis at least 3 times per week .

Exclusion Criteria:

* Receiving nutritional supplementation prior to study commencing or within 1 month of commencement in the study .
* Participants with an allergy to any ingredients in the nutritional supplements.
* Persistent hyperkalemia or hyperphosphatemia (defined as the last 3 months).
* Significant edema and fluid overload.
* Hepatic patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
effect on nutritional status | 3 months
  assessment of nutritional status change at 3 months from baseline using Subjective Global Assessment (SGA)
effect on quality of life | 3 months
  assessment of quality of life change at 3 months from baseline using the kidney disease quality of life 36 (KDQOL-36) short form

SECONDARY OUTCOMES:
effect on BMI | 3 months
  BMI assessment change at 3 months from baseline
mid arm circumference and triceps skin fold | 3 months
  Measurement of mid arm circumference and triceps skin fold change at 3 months from baseline
dialysis adequacy | 3 months
  Estimation of Kt/V change at 3 months from baseline
effect on serum albumin | 3 months
  measurement of serum albumin change at 3 months from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Mamdouh Elsayed, MD, Study Chair — lecturer; Amr El Kazaz, MBBCh, Study Chair — resident; Eman E EL Gohary, MD, Study Chair — Professor; Mohamed M Abdel Kader, MD, Principal Investigator — Professor
Locations (1):
- Faculty of Medicine, Aexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kalantar-Zadeh K, Ikizler TA, Block G, Avram MM, Kopple JD. Malnutrition-inflammation complex syndrome in dialysis patients: causes and consequences. Am J Kidney Dis. 2003 Nov;42(5):864-81. doi: 10.1016/j.ajkd.2003.07.016. PMID 14582032
- [Background] Carrero JJ, Nakashima A, Qureshi AR, Lindholm B, Heimburger O, Barany P, Stenvinkel P. Protein-energy wasting modifies the association of ghrelin with inflammation, leptin, and mortality in hemodialysis patients. Kidney Int. 2011 Apr;79(7):749-56. doi: 10.1038/ki.2010.487. Epub 2010 Dec 22. PMID 21178976
- [Background] Chan M, Kelly J, Batterham M, Tapsell L. Malnutrition (subjective global assessment) scores and serum albumin levels, but not body mass index values, at initiation of dialysis are independent predictors of mortality: a 10-year clinical cohort study. J Ren Nutr. 2012 Nov;22(6):547-57. doi: 10.1053/j.jrn.2011.11.002. Epub 2012 Mar 9. PMID 22406122
- [Background] Ho LC, Wang HH, Peng YS, Chiang CK, Huang JW, Hung KY, Hu FC, Wu KD. Clinical utility of malnutrition-inflammation score in maintenance hemodialysis patients: focus on identifying the best cut-off point. Am J Nephrol. 2008;28(5):840-6. doi: 10.1159/000137684. Epub 2008 Jun 6. PMID 18535370
- [Background] Forquet F, Calin V, Trescol-Biemont MC, Kanellopoulos J, Mottez E, Kourilsky P, Rabourdin-Combe C, Gerlier D. Generation of hen egg lysozyme-specific and major histocompatibility complex class I-restricted cytolytic T lymphocytes: recognition of cytosolic and secreted antigen expressed by transfected cells. Eur J Immunol. 1990 Oct;20(10):2325-32. doi: 10.1002/eji.1830201023. PMID 2242761
- [Derived] Elsayed MM, Abdelkader MM, ElKazaz AM, Elgohary IE. The impact of predialytic oral protein-based supplements on nutritional status and quality of life in hemodialysis patients: a randomized clinical trial. BMC Nephrol. 2025 Feb 26;26(1):103. doi: 10.1186/s12882-025-03999-3. PMID 40011815